CLINICAL TRIAL: NCT00962949
Title: The Renin-Aldosterone Axis in Postural Tachycardia Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Satish R. Raj, Adjunct Assoc Professor, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 081398; PF334
Record Dates: First submitted 2009-08-18; First posted 2009-08-20 (Estimated); Results first posted 2018-08-17 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Postural Orthostatic Tachycardia Syndrome (POTS)
Keywords: POTS; Orthostatic intolerance
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance | interventions — Angiotensin II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Experimental): Healthy controls
  Interventions: Drug: Angiotensin II
- Postural Tachycardia Syndrome (Experimental): Patients with Postural Tachycardia Syndrome
  Interventions: Drug: Angiotensin II

INTERVENTIONS:
Drug: Angiotensin II — Angiotensin II infusion for 1 hour

SUMMARY:
The purpose of this study is to determine the role of the renin-angiotensin-aldosterone in the pathophysiology of postural tachycardia syndrome, and to provide an insight about the disease process in this disorder.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of postural tachycardia syndrome by the Vanderbilt Autonomic Dysfunction Center criteria
* Age between 18-64 years
* Male or females are eligible
* Able and willing to provide informed consent
* Healthy control subjects with no major medical problem (including postural tachycardia syndrome), free of medications during the study

Exclusion Criteria:

* Overt cause of postural tachycardia e.g., dehydration
* Inability to give or withdraw informed consent
* Pregnancy
* Hypertension (BP > 140/90)
* Significant co-morbid condition
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Mustafa HI, Raj SR, Diedrich A, Black BK, Paranjape SY, Dupont WD, Williams GH, Biaggioni I, Robertson D. Altered systemic hemodynamic and baroreflex response to angiotensin II in postural tachycardia syndrome. Circ Arrhythm Electrophysiol. 2012 Feb;5(1):173-80. doi: 10.1161/CIRCEP.111.965343. Epub 2012 Jan 13. PMID 22247480

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Postural Tachycardia Syndrome
Started | 13 | 15
Completed | 13 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Postural Tachycardia Syndrome | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 15 | 28
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Mean Arterial Blood Pressure Change
Description: Change in MAP from baseline to after 1h of infusion.
Time Frame: 1 hour
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Control | Postural Tachycardia Syndrome
Number analyzed (Participants) | 13 | 15
mmHg | 14 (1) | 10 (1)

2. Secondary Outcome: Plasma Renin Activity
Description: Change in plasma renin activity from baseline to after 1h of infusion.
Time Frame: 1 hour
Measure: Mean (Standard Error); unit: micrograms/deciliter
Arm/Group | Control | Postural Tachycardia Syndrome
Number analyzed (Participants) | 13 | 15
micrograms/deciliter | -0.6 (.2) | -0.9 (0.2)

3. Secondary Outcome: Aldosterone Level
Description: Change in aldosterone blood level from baseline to after 1h of infusion.
Time Frame: 1 hour
Measure: Mean (Standard Error); unit: picogram/milliliter
Arm/Group | Control | Postural Tachycardia Syndrome
Number analyzed (Participants) | 13 | 15
picogram/milliliter | 15 (2) | 17 (1)

4. Secondary Outcome: Cortisol Level
Description: Change in cortisol blood level from baseline to after 1h of infusion.
Time Frame: 1 hour
Measure: Mean (Standard Error); unit: ng/ml/h
Arm/Group | Control | Postural Tachycardia Syndrome
Number analyzed (Participants) | 13 | 15
ng/ml/h | -1.4 (0.6) | -0.7 (0.6)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Control | Postural Tachycardia Syndrome
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 0/13 | 0/15

LIMITATIONS AND CAVEATS:
This was a single center, acute study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes